CLINICAL TRIAL: NCT00662896
Title: A 16-week, Phase 1, Multicenter, Double-Blind, Randomized, Naproxen and Ibuprofen-controlled, Parallel-Group Pharmacological Study, to Assess the Effect of Naproxcinod (375mg and750mg, Bid) Compared to Doses of Naproxen (250mg and 500mg, Bid) and to Ibuprofen (600mg, Tid) on Arterial Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring in Osteoarthritis Patients With Controlled Essential Hypertension.
Brief Title: To Assess the Effect of Naproxcinod Versus Naproxen and Ibuprofen on Arterial Blood Pressure in Osteoarthritis Patients With Controlled Essential Hypertension
Acronym: HCT3012-X-112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: NicOx, NicOx.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCT 3012-X-112
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis; Hypertension
MeSH Terms: conditions — Osteoarthritis; Hypertension | interventions — naproxen-n-butyl nitrate; BID protein, human; Naproxen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- naproxcinod 375 mg bid (Experimental)
  Interventions: Drug: naproxcinod 375 mg bid
- naproxen 250 mg bid (Active Comparator)
  Interventions: Drug: naproxen 250 mg bid
- ibuprofen 600 mg tid (Active Comparator)
  Interventions: Drug: ibuprofen 600 mg tid
- naproxcinod 750 mg bid (Experimental)
  Interventions: Drug: naproxcinod 750 mg bid
- naproxen 500 mg bid (Active Comparator)
  Interventions: Drug: naproxen 500 mg bid

INTERVENTIONS:
Drug: naproxcinod 375 mg bid — naproxcinod 375 mg bid
  Arms: naproxcinod 375 mg bid
Drug: naproxcinod 750 mg bid — naproxcinod 750 mg bid
  Arms: naproxcinod 750 mg bid
Drug: naproxen 250 mg bid — naproxen 250 mg bid
  Arms: naproxen 250 mg bid
Drug: naproxen 500 mg bid — naproxen 500 mg bid
  Arms: naproxen 500 mg bid
Drug: ibuprofen 600 mg tid — ibuprofen 600 mg tid
  Arms: ibuprofen 600 mg tid

SUMMARY:
To assess the effect of naproxcinod vs. naproxen and ibuprofen on arterial blood pressure in patients with osteoarthritis and controlled essential hypertension

DETAILED DESCRIPTION:
This is a 16-week, randomized, double-blind, multicenter study comparing the effect of naproxcinod, naproxen, and ibuprofen on 24 hour arterial blood pressure profile. Patients will be randomly allocated to naproxcinod 375mg, naproxcinod 750mg, naproxen 250mg, naproxen 500mg, or ibuprofen 600mg in a 1:1:1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women, 40 or older, diagnosed with hip or knee osteoarthritis.
* Hypertensive Patient with treated and controlled essential hypertension.
* Must receive at least one antihypertensive treatment from the following drug classes: Diuretic, Angiotensin-Converting Enzyme (ACE) inhibitor, Angiotensin Receptor Blockers (ARB) or Beta-Blocker (BB).
* Must be current chronic user of NSAIDS or acetaminophen.
* Must discontinue all analgesic therapy at Screening.

Exclusion Criteria:

* More than two different classes of antihypertensive drugs.
* Uncontrolled diabetes.
* Hepatic or renal impairment.
* A history of alcohol/drug abuse.
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding.
* History of congestive heart failure.
* Clinically relevant abnormal ECG.
* Current or history of a medical disease that could interfere with the study objectives or put the patient's safety at risk.
* Current or expected use of anticoagulants.
* Participation within 30 days prior to pre-screening in another investigational study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To characterize the 24-hour arterial blood pressure profile of naproxcinod, compared to naproxen as measured by ABPM, through assessing the mean change from baseline in patients with OA and controlled essential hypertension. | 15 weeks

SECONDARY OUTCOMES:
To characterize the 24-hour arterial blood pressure profile of naproxcinod compared to ibuprofen as measured by ABPM, through assessing the mean change from baseline in patients with osteoarthritis and controlled essential hypertension. | 15 weeks
To assess the general safety and tolerability of naproxcinod compared to naproxen and ibuprofen. | 15 weeks

CONTACTS AND LOCATIONS:
Locations (57):
- United States (57):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Sierra Vista, Arizona
  - Carmichael, California
  - Fair Oaks, California
  - Long Beach, California
  - Pico Rivera, California
  - Upland, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Milford, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Arlington Heights, Illinois
  - Peoria, Illinois
  - Elizabethtown, Kentucky
  - Erlanger, Kentucky
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - Towson, Maryland
  - Florissant, Missouri
  - Missoula, Montana
  - Grand Island, Nebraska
  - Henderson, Nevada
  - Albuquerque, New Mexico
  - Rochester, New York
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Hickory, North Carolina
  - Lenoir, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Havertown, Pennsylvania
  - Tipton, Pennsylvania
  - Charleston, South Carolina
  - Kingsport, Tennessee
  - New Tazewell, Tennessee
  - Dallas, Texas
  - Irving, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin

REFERENCES:
- See also: Nicox web-site — http://www.nicox.com